CLINICAL TRIAL: NCT04579718
Title: A Multicenter Study on the Feasibility of a Radiotherapy Treatment Planning System (TPS) Software---Zeus Cloud
Brief Title: A Study of Radiotherapy Planning System Software ---- Zeus Cloud
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); The Affilicated Suzhou Science and Technology Town Hospital (Unknown)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Other Study IDs: GASTO-1062
Record Dates: First submitted 2020-09-26; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Radiotherapy
Keywords: Treatment Planning System
MeSH Terms: interventions — Eclipse Prosthodontic Resin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eclipse
  Interventions: Other: Eclipse
- Zeus Cloud TPS V1.0
  Interventions: Other: Zeus Cloud TPS V1.0

INTERVENTIONS:
Other: Zeus Cloud TPS V1.0 — Zeus Cloud TPS V1.0 is used to design the radiotherapy plan for the subjects and the plan is evaluated.
  Groups: Zeus Cloud TPS V1.0
Other: Eclipse — Eclipse TPS of Varian company is used to design the radiotherapy plan for the subjects and the plan is evaluated.
  Groups: Eclipse

SUMMARY:
To evaluate the feasibility of Zeus Cloud TPS in the design of photon intensity modulated radiation therapy (IMRT) plan for tumors in various parts of the body.

DETAILED DESCRIPTION:
This is a self-control, multi-center non-inferiority study. Subjects meeting inclusion criteria have radiation treatment plans designed by Zeus Cloud TPS and Eclipse treatment planning software from Varian, respectively. The qualities of two plans are compared.

This is a observational study as the two plans are not executed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed brain glioma, nasopharyngeal carcinoma, lung cancer, esophageal cancer, gastric cancer, liver cancer, prostate cancer, cervical cancer and rectal cancer;
2. The medical imaging data (CT) of the subjects were complete and available;
3. Between 18 and 75 years old, regardless of gender;

Exclusion Criteria:

1. The patients had metal implants;
2. Not suitable for clinical trials judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed brain glioma, nasopharyngeal carcinoma, lung cancer, esophageal cancer, gastric cancer, liver cancer, prostate cancer, cervical cancer and rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
The qualification rate of treatment plans based on dosimetry | 2 months

SECONDARY OUTCOMES:
The conformability index of radiation dose to the target | 2 months
single-field pass rate | 2 months
composite-field pass rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Prof., Principal Investigator — Sun Yat-sen University